CLINICAL TRIAL: NCT06633900
Title: Extended-Release Naltrexone as Opioid Overdose Pre-Exposure Prophylaxis (PrEP) in People Using Stimulants Living With or At Risk of HIV
Brief Title: Naltrexone for Overdose Prevention
Acronym: NOD
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 24-41278; 1DP2DA060600-01 (NIH)
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Overdose Accidental
Keywords: stimulants; cocaine; methamphetamine; overdose prevention; naltrexone; fentanyl exposure

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either receive the study medication or usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants assigned to the intervention arm will receive naltrexone injections once a month over 6 months. The naltrexone injection (380mg) will be administered every 4 weeks in the ventrogluteal location.
  Interventions: Drug: IM naltrexone
- Control (Active Comparator): Participants in the control arm will receive usual care.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Drug: IM naltrexone — The study drug is an intramuscular injection of naltrexone (380mg), administered every 4 weeks via an injection in the ventrogluteal region.
  Arms: Intervention
Behavioral: Usual Care — Participants assigned to usual care will receive a harm reduction bundle in clinic. It will include the following components: 1) intranasal naloxone 4mg x 2, 2) participant choice of safer consumption kits based on substances and route used (specific materials for inhaled use vs. injecting, based on common use practices in the region), 3) fentanyl test kits with 2 lateral flow assays per package along with instructions to minimize false positive results, and 4) information about universal overdose precautions (behavioral modifications to optimize safety like using in the presence of others, use a test dose of new substances, etc.)
  Arms: Control

SUMMARY:
The goal of this clinical trial is to see if an injectable medicine called naltrexone can prevent fentanyl overdose deaths in people who use other drugs (cocaine, methamphetamine). The main questions it aims to answer are:

What are the challenges for implementing naltrexone as an overdose prevention strategy?

Are injections of naltrexone effective for opioid overdose prevention among people who use stimulants?

How often are people who use stimulants and do not intentionally use opioids unintentionally exposed to opioids?

Researchers will compare participants to receive the study medication to the usual care group to see if one group experiences fewer opioid overdose events than the other.

Participants will be randomized to either receive a monthly injection of naltrexone over six months, or receive usual care. Usual care includes harm reduction supplies. Laboratory procedures will include the collection of urine, blood, and hair samples for various safety and outcome measure testing.

DETAILED DESCRIPTION:
This pilot randomized controlled trial aims to evaluate the efficacy of IM naltrexone for opioid overdose prevention among individuals living with HIV (PWH) and those at risk for HIV who use stimulants. The study will concurrently collect data on the feasibility, acceptability, and preliminary effectiveness of the intervention, along with epidemiological data on the prevalence of both intentional and unintentional fentanyl exposure in this population.

Participants will be randomly assigned in a 1:1 fashion to either the intervention group, which will receive IM naltrexone, or the usual care group, which will be provided with safe consumption supplies and intranasal naloxone.

Monthly assessments over a 24-week period post-intake (followed by a final study visit at 32 weeks) will be conducted to measure participants' exposure to fentanyl/opioids, utilizing both short-term (urine) and long-term (hair) biomarkers, as well as self-reported data. Adherence to the monthly IM naltrexone injections and the safety profile of the 'opioid PrEP' will also be rigorously evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. at-risk for HIV or living with HIV
2. stimulant use disorder (by DSM-V) or positive urine drug test for cocaine, amphetamine, or methamphetamine in last 6 months AND report at least 10 days of stimulant use/month,
3. able to provide informed consent,
4. English-speaking,
5. age 18 years old or greater.

Exclusion Criteria:

1. prescribed or non-prescribed opioid use (including newly diagnosed opioid use disorder by DSM-V),
2. receipt of long-acting injectable naltrexone for other indications in past 30 days,
3. planned surgery in next 6 months,
4. moderate, severe or chronic liver disease (AST, ALT ≥ 5 times the upper limit of normal or symptoms of current liver disease),
5. persons who are pregnant or breastfeeding,
6. increased risk of bleeding (thrombocytopenia <50 x 109/L, coagulopathy, or therapeutic anticoagulation), or
7. known hypersensitivity to naltrexone or its diluents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 6 months
  The primary outcome is the acceptability of IM naltrexone as opioid PrEP, which the study investigators will quantitatively assess via retention in treatment at 24 weeks and proportion of on-time injections during the study period. The investigators will consider 50% of enrolled participants completing 3 or more injections to meet a minimum standard of intervention uptake.

SECONDARY OUTCOMES:
Effectiveness | 6 months
  The study investigators will also evaluate incident opioid overdose, which will be defined as 1) fatal overdose, 2) overdose requiring emergency medical services (including first-responder evaluation, emergency department visit, hospitalization), or 3) participant report of overdose or sedation responding to community-delivered naloxone. This will allow the investigators to define unintentional opioid overdose rates among PWH or individuals at risk only seeking to use stimulants (with inadvertent exposure to opioids) while also evaluating possible effectiveness of IM naltrexone as an augmented harm reduction strategy.
Safety | 6 months
  Our primary safety outcome is proportion of participants with grade 2 or worse adverse events (such as nausea, vomiting, laboratory abnormalities, neurologic symptoms).

OTHER OUTCOMES:
Opioid exposure | 6 months
  As an additional biomarker-based method of evaluating possible opioid overdose prevention, the investigators will analyze participant hair for opioids and compare this to the measure of opioid overdose during the same time period. Hair samples can be analyzed for opioids or methamphetamines as a cumulative metric of exposure. If a participant on IM naltrexone is found to have fentanyl-positive hair (indicating exposure in the last 1-3 months depending on length analyzed) but no clinical overdose, this may suggest an unrecognized exposure, and possible protection by naltrexone. Hair can also be used to evaluate temporal trends in stimulant use quantity to record reduced use in the intervention arm vs. usual care arm.
Viral suppression | 6 months
  HIV viral suppression will be recorded at baseline and time of exit from the trial to evaluate whether increased engagement in clinic-based harm reduction efforts has a positive effect upon successful HIV control.

CONTACTS AND LOCATIONS:
Overall Officials: Ayesha Appa, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Center on Substance Use and Health, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No